CLINICAL TRIAL: NCT07176130
Title: Demographics and Clinical Characteristics of Ocular Inflammatory Diseases in Singapore
Status: Active, not recruiting | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Samanthila Waduthantri, Principal Resident Physician, Singapore National Eye Centre
Other Study IDs: 2019/2811
Record Dates: First submitted 2025-08-30; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Uveitis; Scleritis and Episcleritis; Endophthalmitis; Masquerade Syndromes; Intraocular Lymphoma
Keywords: Uveitis; Scleritis; Masquerades syndromes; Intraocular lymphoma; Endophthalmitis
MeSH Terms: conditions — Uveitis; Scleritis; Endophthalmitis; Intraocular Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Uveitis: Patients diagnosed with uveitis at Singapore National Eye Centre
  Interventions: Other: No Intervention: Observational Cohort
- Scleritis and Episcleritis: Patients diagnosed with scleritis or episcleritis at Singapore National Eye Centre
  Interventions: Other: No Intervention: Observational Cohort
- Intraocular lymphoma: Patients diagnosed with ocular neoplasms at Singapore National Eye Centre
  Interventions: Other: No Intervention: Observational Cohort
- Endophthalmitis: Patients diagnosed with endophthalmitis at Singapore National Eye Centre
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — Not applicable, No intervention. Observational study.

SUMMARY:
This is a retrospective study analyzing demographics, clinical characteristics, treatment received, and outcomes of ocular inflammatory diseases that presented to the Singapore National Eye Centre (SNEC).

DETAILED DESCRIPTION:
This is a retrospective, cross-sectional study. In this study, the investigators aim to investigate demographics, clinical characteristics, treatment received, and outcomes of ocular inflammatory diseases, including masquerade syndromes such as ocular neoplasms (e.g., vitreoretinal and uveal lymphoma) and endophthalmitis that presented to the Singapore National Eye Centre (SNEC). Data on demographics, clinical features, diagnosis, investigations, secondary complications, treatment received, and outcomes will be analyzed using statistical software. The results of this study will lead to an improved clinical practice with better treatment selections and an optimized monitoring protocol for follow-up care for patients with ocular inflammatory diseases, including masquerade syndromes such as ocular neoplasms (e.g.,vitreoretinal and uveal lymphoma) and endophthalmitis. This will lead to better clinical outcomes and prevention of serious sight-threatening complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with uveitis
* Patients diagnosed with scleritis or episcleritis
* Patients diagnosed with ocular neoplasms e.g., vitreoretinal and uveal lymphoma
* Patients diagnosed with endophthalmitis
* Diagnosis confirmed by laboratory testing or histopathological examination
* Patients diagnosed and managed at the Singapore National Eye Centre (SNEC)

Exclusion Criteria:

* Patients with less than two years of clinical follow-up
* Patients with incomplete diagnostic confirmation (i.e., lacking laboratory or histopathological evidence)
* Patients diagnosed outside of Singapore National Eye Centre (SNEC)
* Cases with missing key clinical or outcome data

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with ocular inflammatory diseases, including masquerade syndromes such as ocular neoplasms (e.g., vitreoretinal and uveal lymphoma) and endophthalmitis, at the Singapore National Eye Centre.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Distribution of demographics, diagnosis, clinical features, treatment and outcomes | January 1987 and January 2025
  Percentage ethnic distribution, percentage of gender distribution, percentage of age distribution, percentage of etiology, percentage of clinical features, percentage of investigations, percentage of diagnosis, percentage of secondary complications, percentage of treatment received, percentage of outcomes

SECONDARY OUTCOMES:
Correlation of demographics, diagnosis, clinical features, and treatment outcomes | January 1987 and January 2025
  To evaluate the independent and combined effects of demographic factors, diagnostic categories, and clinical features on treatment outcomes using multivariate logistic and cox regression analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. Anonymous data.

REFERENCES:
- [Background] Siak J, Jansen A, Waduthantri S, Teoh CS, Jap A, Chee SP. The Pattern of Uveitis among Chinese, Malays, and Indians in Singapore. Ocul Immunol Inflamm. 2017;25(sup1):S81-S93. doi: 10.1080/09273948.2016.1188968. Epub 2016 Jul 15. PMID 27419535
- [Background] Chee SP, Jap A. Endogenous endophthalmitis. Curr Opin Ophthalmol. 2001 Dec;12(6):464-70. doi: 10.1097/00055735-200112000-00012. PMID 11734687
- [Background] International Vitreoretinal B-Cell Lymphoma Registry Investigator Group. Presentation, Diagnostic Testing and Initial Treatment of Vitreoretinal Lymphoma. Ophthalmol Retina. 2024 Jan;8(1):72-80. doi: 10.1016/j.oret.2023.08.012. Epub 2023 Aug 28. PMID 37648063
- [Background] Carbonell D, Mahajan S, Chee SP, Sobolewska B, Agrawal R, Bulow T, Gupta V, Jones NP, Accorinti M, Agarwal M, Batchelor T, Biswas J, Cimino L, tenDam-van Loon NH, de-la-Torre A, Frenkel S, Pe'er J, Kramer M, Miserocchi E, Mochizuki M, Ness T, Rosenbaum JT, Sen HN, Simion M (VRL patient), Sitter H, Vasconcelos-Santos DV, Habot-Wilner Z, Coupland SE, Pulido JS, Smith J, Thorne JE, Zierhut M; Study Group for Vitreoretinal Lymphoma Diagnostics. Consensus Recommendations for the Diagnosis of Vitreoretinal Lymphoma. Ocul Immunol Inflamm. 2021 Apr 3;29(3):507-520. doi: 10.1080/09273948.2021.1878233. Epub 2021 May 19. PMID 34009095